CLINICAL TRIAL: NCT02721940
Title: Local Administration of Enriched Mononuclear Cells, Platelets and Zoledronic Acid for Preventing Collapse of the Femoral Head in the Early Stage of Osteonecrosis: a Prospective, Randomized, Parallel-controlled Clinical Trial
Brief Title: Mononuclear Cells, Platelets and Zoledronic Acid for Preventing Collapse of the Femoral Head in Osteonecrosis
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Chinese PLA General Hospital (Other)
Responsible Party: Principal Investigator, Quanyi Guo, Director, Chinese PLA General Hospital
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: PLAGH_001
Record Dates: First submitted 2016-03-17; First posted 2016-03-29 (Estimated); Last update posted 2016-03-29 (Estimated); Status verified 2016-03

CONDITIONS: Osteonecrosis
MeSH Terms: conditions — Osteonecrosis | interventions — Control Groups; Platelet Count; Zoledronic Acid; Saline Solution

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Treatment group (Experimental): In the treatment group, patients will be given local injection of enriched autologous mononuclear cells and zoledronic acid into the necrotic area following core decompression by drilling.
  Interventions: Biological: Mononuclear Cells; Biological: Platelets; Drug: Zoledronic Acid; Drug: Normal saline
- Control group (Experimental): In the control group, core decompression will be performed, but no treatment will be given.
  Interventions: Procedure: Control group

INTERVENTIONS:
Procedure: Control group — Patients in the control group will be subjected to arthroscopic debridement and microfracture surgery.
  Other Names: Arthroscopic debridement and microfracture surgery
  Arms: Control group
Biological: Mononuclear Cells — In the treatment group, patients will be given 200 μg zoledronic acid and purified bone marrow mononuclear cells will be injected into the necrotic zone, followed by injection of 5-10 mL normal saline. Finally, the holes for core decompression will be sealed with a small amount of bone wax to prevent leakage.
  Arms: Treatment group
Biological: Platelets — In the treatment group, patients will be given 200 μg zoledronic acid and purified bone marrow mononuclear cells will be injected into the necrotic zone, followed by injection of 5-10 mL normal saline. Finally, the holes for core decompression will be sealed with a small amount of bone wax to prevent leakage.
  Arms: Treatment group
Drug: Zoledronic Acid — In the treatment group, patients will be given 200 μg zoledronic acid and purified bone marrow mononuclear cells will be injected into the necrotic zone, followed by injection of 5-10 mL normal saline. Finally, the holes for core decompression will be sealed with a small amount of bone wax to prevent leakage.
  Arms: Treatment group
Drug: Normal saline — In the treatment group, patients will be given 200 μg zoledronic acid and purified bone marrow mononuclear cells will be injected into the necrotic zone, followed by injection of 5-10 mL normal saline. Finally, the holes for core decompression will be sealed with a small amount of bone wax to prevent leakage.
  Arms: Treatment group

SUMMARY:
This study was mainly aimed to evaluate the efficacy of local administration of enriched bone marrow mononuclear cells, platelets and zoledronic acid for the clinical prevention of collapse of the early-stage osteonecrotic femoral head.

DETAILED DESCRIPTION:
Osteonecrosis of the femoral head (ONFH) is a common degenerative disease caused by a variety of factors, such as trauma, alcoholism, use of corticosteroids, and systemic lupus erythematosus. In ONFH, the overall mechanical properties of the femoral head change over time, and collapse of the femoral head results in severe pain and disability.

Although there are numerous strategies for treating ONFH, conservative treatments are often ineffective. Once collapse of the femoral head occurs, hip replacement is the only option for ONFH patients. Therefore, it is important to reduce osteonecrotic weakening of the femoral head in the early stage of ONFH to prevent subsequent head collapse. Studies have shown that bisphosphonates inhibit osteoclast activity, reduce bone resorption, retain bone trabeculae, reduce apoptosis of osteoblasts and osteocytes, and promote new bone formation. Therefore, investigators have chosen to use bisphosphonates for preventing collapse of the osteonecrotic femoral head. Zoledronic acid is the most potent bisphosphonate for the treatment of ONFH. It can reduce bone resorption and preserve the shape of the femoral head. In most cases, bisphosphonates are given intravenously or orally. However, systemic administration is associated with many complications, including osteonecrosis of the mandible and atypical femur fractures. As previously reported, poly(lactic-co-glycolic acid) acts as a drug carrier to facilitate the local release of zoledronic acid, and it has been found to promote bone formation and help avoid the complications caused by systemic administration. Using this method of administration, zoledronic acid can reach locally therapeutic levels, thereby preventing femoral head collapse.

ONFH reduces the viability of bone marrow hematopoietic cells and bone cells to varying degrees, and can even induce cell death. Adult red bone marrow has two distinct parts; a hematopoietic section containing hematopoietic stem cells, and a mesenchymal section containing mesenchymal stem cells that promote bone regeneration. Core decompression technology can reduce intraosseous pressure, improve venous return, promote revascularization of the femoral head, and effectively reduce the symptoms of osteonecrosis; however, clinical efficacy is currently unsatisfactory, probably because of insufficient bone formation and repair. In recent years, the use of bone marrow mononuclear cells (BMMCs) has shown good short-term clinical efficacy in the treatment of ONFH. However, the long-term outcome is unknown, and it is not known whether combined therapy with platelet-rich plasma may be effective for the treatment of femoral head collapse in the early stage of ONFH.

Here, investigators propose a prospective, randomized controlled trial to assess the clinical efficacy of local administration of enriched BMMCs, platelets and zoledronic acid for preventing femoral head collapse in the early stage of ONFH.

Safety assessment During the trial, inspectors will be responsible for monitoring adverse reactions in the patients. If any adverse reaction is observed during the follow-up, the patient will be urged to call their doctor for assistance. Predicted complications include fever, joint pain, joint snapping, joint noise, joint swelling, limited mobility, and itchy skin. Patients will be urged to inform their family members or close friends to observe for these symptoms and that they are participating in a clinical trial. If a patient has questions about participating in this trial, they will be informed how to contact their doctor. All serious adverse events will be recorded in detail-including the date of occurrence, duration, treatments, and possible relationships with the therapeutic procedures-and reported to the research director and the ethics committee within 24 hours.

Data collection and management All the data will be collected on a case report form, including demographic information, disease diagnosis, and concomitant diseases. Data will be recorded electronically using a double-data entry strategy. After the follow-up, all the data will be checked and locked by the principal investigator. The locked data, which cannot be modified, will be saved for subsequent analysis. All the data relevant to this clinical trial will be saved by the Chinese PLA General Hospital. Then, the data will be statistically analyzed by professional statisticians, and the statistical results will be reported to the principle investigator who will be responsible for writing the research report. The Data Monitoring Committee (IDMC) will be responsible for data monitoring and management throughout the entire trial, to ensure scientific accuracy, authenticity, and integrity.

Statistical analysis Data will be statistically analyzed using SPSS 22.0 (IBM, Armonk, NY, USA). Measurement data that are normally distributed will be expressed as mean, standard deviation, minimum value and maximum value. Data that are non-normally distributed will be expressed as the lower quartile (q1), median and upper quartile (q3). Count data will be expressed as a percentage (%).

Where appropriate, two-tailed tests will be used, with statistical significance set at P < 0.05. Baseline data will be compared between groups, and statistically analyzed using two-tailed tests at α = 0.05. Count data will be compared between groups using chi-square test or Fisher exact test. Measurement data will be compared between groups using t-tests, and nonparametric variables will be compared between groups using the rank sum test.

ELIGIBILITY:
Inclusion Criteria:

* 14-55 years of age
* Either sex
* Patients with Ficat I-II ONFH confirmed by anteroposterior and lateral X-ray and CT films
* No collapse of the femoral head
* No previous ONFH-related surgery
* Tolerant to anesthesia and surgical procedures

Exclusion Criteria:

* Inability to tolerate surgical procedures
* Blood diseases
* Bleeding tendency
* Drug addictions (narcotics, anesthetics and/or alcohol)
* Inflammatory arthritis (specific or non-specific arthritis)
* Immune system disorders
* Metabolic disease (gout, rheumatism)
* Lactating or pregnant women, or women who are preparing to conceive within

  1 year after initial recruitment
* Patients with psychiatric disorders who have poor compliance and cannot complete the rehabilitation therapy

Ages: 14 Years to 55 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 100 (Actual)
Dates: Start 2012-02; Primary Completion 2015-01 (Actual); Study Completion 2016-05 (Estimated)

PRIMARY OUTCOMES:
Change of Magnetic resonance imaging(MRI) | Before treatment and month 3, month 6, month 12,month 18 after surgery
  Dynamic perfusion MRI to observe the blood supply in the necrotic area

SECONDARY OUTCOMES:
Change of Three-dimensional CT | Before treatment and month 3, month 6, month 12,month 18 after surgery
  Three-dimensional CT reconstruction of the hip joint to observe new bone formation in the necrotic area
Change of X-ray film | Before treatment and month 3, month 6, month 12,month 18 after surgery
  Anteroposterior and lateral X-ray films to observe the outline of the femoral head
Change of Harris score | Before treatment and month 3, month 6, month 12,month 18 after surgery
  Harris score of the hip joint to assess hip joint function
Change of Numerical rating scale(NRS) score | Before treatment and month 3, month 6, month 12,month 18 after surgery
Change of SF-36 score | Before treatment and month 3, month 6, month 12,month 18 after surgery
Change of Activities of Daily Living (ADL) score | Before treatment and month 3, month 6, month 12,month 18 after surgery

CONTACTS AND LOCATIONS:
Overall Officials: Quanyi Guo, Ph.D, Principal Investigator — Institute of Orthopedics, Chinese PLA Hospital, Beijing, China

IPD SHARING:
Plan to Share IPD: Undecided